CLINICAL TRIAL: NCT01277874
Title: Oscillatory Versus Non-Oscillatory Nasal Continuous Airway Pressure Neonatal Respiratory Support
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI has left Institution
Sponsor: University of Utah (Other)
Responsible Party: Donald Null M.D., University of Utah / Primary Childrens Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36738
Record Dates: First submitted 2011-01-13; First posted 2011-01-17 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Respiratory Distress Syndrome; Prematurity
MeSH Terms: conditions — Respiratory Distress Syndrome; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nasal CPAP (Active Comparator): Standard Nasal CPAP
  Interventions: Device: Nasal CPAP
- Oscillatory NCPAP (Active Comparator): NCPAP will be given to infant via prongs in the infant's nose. A Bird Industries pneumatic oscillating diaphragm to drive a Bird Industries phasatron which is attached by T-connector to the NCPAP patient circuit.
  Interventions: Device: Oscillatory NCPAP

INTERVENTIONS:
Device: Nasal CPAP — NCPAP is delivered via nasal prongs placed into infant's nares. It may be delivered via ventilator or by bubble.
  Arms: Nasal CPAP
Device: Oscillatory NCPAP — Bird Industries pneumatic diaphragm is attached to NCPAP patient circuit to provide oscillations.
  Other Names: Bird Industries
  Arms: Oscillatory NCPAP

SUMMARY:
This study will seek to enroll neonates requiring Nasal Continuous Airway Pressure (NCPAP) respiratory support and randomize them to either oscillatory (Osc-NCPAP, study group) or non-oscillatory (NCPAP, control group) mode. The goal of the research is to determine if Osc-NCPAP provides improved ventilation support compared to routine NCPAP, i.e. NCPAP without oscillations. This will be measured by need for change to ventilator support, improvement in pCO2 values, and reduction in respiratory rate and frequency of apnea during the period of NCPAP treatment. Other respiratory outcomes will also be compared, including time on NCPAP, time on High-Flow Nasal Cannula support following NCPAP, and time-averaged PiO2 from start of study to end of respiratory treatment.

ELIGIBILITY:
Inclusion Criteria:

* Newborn (0-28 days of age) admitted to Neonatal Intensive Care Unit (NICU)
* Ordered respiratory treatment of NCPAP

Exclusion Criteria:

* Major congenital defect
* Known or suspected chromosomal disorder

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Physiologic respiratory stability of Oscillating versus Non-Oscillating NCPAP | 2 months
  Determine the physiologic respiratory stability (pCO2, respiratory rate, apnea frequency) during treatment with NCPAP
Need for mechanical ventilation following the initiation of NCPAP. | 2 months
  The rate of mechanical ventilation following both Oscillating and Non-Oscillating groups.

SECONDARY OUTCOMES:
Total duration of non-invasive and invasive respiratory support in each study group. | 2 months
  Determine the total duration of non-invasive and invasive respiratory support in each study group.
total amount of oxygen exposure in each study group. Total amount of oxygen exposure in each study group. | 2 months
  Determine the total amount of oxygen exposure in each study group.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Null, MD, Principal Investigator — University of Utah
Locations (3):
- United States (3):
  - Valley Children's Healthcare, Madera, California
  - Primary Children's Medical Center, Salt Lake City, Utah
  - University of Utah Health Sciences Center, Salt Lake City, Utah